CLINICAL TRIAL: NCT01142999
Title: Feasibility Study of Barrier Enhancement for Eczema Prevention (BEEP)
Brief Title: Feasibility Study of Barrier Enhancement for Eczema Prevention
Acronym: BEEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Eric L. Simpson, M.D., M.C.R., Oregon Health & Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BEEP
Record Dates: First submitted 2010-06-10; First posted 2010-06-14 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2010-06

CONDITIONS: Eczema
MeSH Terms: conditions — Eczema | interventions — Sunflower Oil; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (moisturizer group) (Active Comparator): One group will be instructed to use a choice of 3 FDA-approved moisturizers and soap substitutes on their newborn infants.
  Interventions: Drug: Sunflower oil; Drug: Aquaphor ointment; Drug: Cetaphil cream
- Control group (no moisturizers) (Active Comparator): This group will be asked NOT to use any skin moisturizers and use only soap substitutes on their infants.
  Interventions: Drug: Control group

INTERVENTIONS:
Drug: Sunflower oil — One group will be instructed to use FDA-approved moisturizers and soap substitutes on their newborn infants.
  Other Names: Moisturizers
  Arms: Intervention (moisturizer group)
Drug: Control group — This group will be asked NOT to use any skin moisturizers and use only soap substitutes on their infants.
  Arms: Control group (no moisturizers)
Drug: Aquaphor ointment — One group will be instructed to use FDA-approved moisturizers and soap substitutes on their newborn infants.
  Arms: Intervention (moisturizer group)
Drug: Cetaphil cream — One group will be instructed to use FDA-approved moisturizers and soap substitutes on their newborn infants.
  Arms: Intervention (moisturizer group)

SUMMARY:
The purpose of this protocol is to determine the feasibility of doing larger follow-up studies examining whether emollients used from birth can prevent eczema in high-risk babies and to help investigators find out if emollients (moisturizing skin creams) used from birth can prevent eczema in high-risk babies. Hypothesis: Enhancing the skin barrier from birth using emollients will prevent or delay the onset of eczema, especially in predisposed infants.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have a parent or sibling with a history of at least one of the following: eczema, allergic rhinitis or asthma
2. Infant in overall good health
3. Mother between the ages of 16 and 45 years of age at delivery; infant from birth thru 6 months of age
4. Capable of giving informed consent

Exclusion Criteria:

1. Preterm birth defined as birth prior to 37 weeks gestation
2. Major congenital anomaly
3. Hydrops fetalis
4. Significant dermatitis at birth not including seborrheic dermatitis ("cradle cap")
5. Any immunodeficiency disorder or severe genetic skin disorder
6. Any other serious condition that would make the use of emollients inadvisable
7. Any other major medical problems that the investigator deems may increase the risk of adverse events with the intervention

Ages: 1 Minute to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2010-05; Primary Completion 2011-08 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of families willing to be randomized. | 6 months
  Determine proportion of families willing to be randomized in order to design larger study in the future.

SECONDARY OUTCOMES:
Proportion of families eligible for the trial, willing to participate | 6 months
Proportion of families who found the interventions acceptable | 6 months
Reported adherence with intervention | 6 months
Proportion of families for whom the blinding of the assessor to the allocation ostatus was not compromised | 6 months
Amount of contamination as a result of increased awareness in the control group | 6 months
Percentage of missing data and early withdrawal rates | 6 months
Incidence of emollient-related adverse events | 6 months
Incidence of eczema at 6 and 12 months | 12 months
Age at onset of eczema | 6 months
Filaggrin mutation status | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric L. Simpson, M.D., M.C.R., Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States